CLINICAL TRIAL: NCT04814849
Title: Long-term Occupational Consequences for Families of Children With Type 1 Diabetes: the Mothers Take the Burden
Brief Title: Parents' Occupation After Diabetes Onset
Acronym: AMBA
Status: Completed | Type: Observational
Sponsor: Hannover Medical School (Other)
Collaborators: diabetesDE-Deutsche Diabetes Hilfe (Unknown); Sana-Klinikum Lichtenberg (Other); Kinderkrankenhaus auf der Bult (Other); Katholisches Kinderkrankenhaus Wilhelmstift (Unknown); Evangelisches Krankenhaus Bielefeld gGmbH (Other); Elisabeth-Krankenhaus Essen (Unknown); Ruhr University of Bochum (Other); Leopoldina-Krankenhaus der Stadt Schweinfurt GmbH (Unknown); Kinderärzte Mondstraße, Dr. med. Ralph Ziegler und Kollegen, Praxis für Kinder und Jugendmedizin (Unknown)
Responsible Party: Principal Investigator, Heike Saßmann, Dr., Dr. Heike Saßmann, Hannover Medical School
Other Study IDs: 260320597
Record Dates: First submitted 2021-03-18; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes, parents, occupation, gender inequality
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A cross-sectional multicenter study using a questionnaire assessing occupational and financial situation before and after the onset of type 1 diabetes was distributed to all families with a child diagnosed with type 1 diabetes before the age of 14 years in nine German pediatric diabetes centers.

DETAILED DESCRIPTION:
This cross-sectional multicenter study was conducted between January and June 2018 during a three months period per center. The selected nine pediatric diabetes centers covered all regions of Germany. The study participants were mothers, fathers, or other primary caregivers of children and adolescents diagnosed with type 1 diabetes before 14 years of age. During a regularly scheduled medical visit, in Germany usually 4 per year, families were informed about the study procedure, its aims and anonymous data collection and analyses. The answered questionnaires were either collected in a closed box in each diabetes center or could be sent anonymously via a prepaid envelope to the study administration center.

ELIGIBILITY:
Inclusion Criteria:

* mothers, fathers or other primary caregivers of children and adolescents diagnosed with type 1 diabetes before 14 years of age
* child's diabetes duration at least 12 months
* child's age under 19 years

Exclusion Criteria:

* caregivers unability to understand German language sufficiently

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Of 1470 eligible families in the nine centers, 1192 (81% response rate) agreed to participate and answered the questionnaire. The majority of respondents to the questionnaire were mothers (n = 939; 82%). Overall 48 questionnaires had to be excluded due to a high number of missing data. Thus, the final sample consisted of n = 1144 answered questionnaires with information about both parents' occupational situation.
Sampling Method: Non-Probability Sample
Enrollment: 1144 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
occupational situation of parents | up to 12 weeks
  questionnaire with 7 items to capture changes in occupational situation of parents after the onset of type 1 diabetes in their child
number of participants reporting financial burden | up to 12 weeks
  questionnaire to capture changes in occupational situation of parents after the onset of type 1 diabetes in their child

SECONDARY OUTCOMES:
number of participants reporting emotional and/or psychosocial burden | up to 12 weeks
  questionnaire to capture psychosocial and emotional burden of parents in the year following the diagnosis of diabetes in a child

CONTACTS AND LOCATIONS:
Overall Officials: Karin Lange, PhD, Study Director — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No